CLINICAL TRIAL: NCT00995345
Title: A 24-Week, Randomized, Double-Blind, Placebo-Controlled Study to Asses the Safety and Efficacy of Once-Daily KRP-104 in Patients With Type 2 Diabetes With Inadequate Glycemic Control on Metformin Alone.
Brief Title: Safety and Efficacy of Once-Daily KRP-104 in Type 2 Diabetics With Inadequate Glycemic Control on Metformin Alone
Acronym: Synergy104
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ActivX Biosciences, Inc. (Industry)
Collaborators: Kyorin Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0104-005
Record Dates: First submitted 2009-10-12; First posted 2009-10-15 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose 1: KRP-104 40 mg (Experimental): Tablet, once-daily for 24 weeks
  Interventions: Drug: KRP-104
- Dose 2: KRP-104 80 mg (Experimental): Tablet, once-daily for 24 weeks
  Interventions: Drug: KRP-104
- Dose 3: KRP-104 100 mg (Experimental): Tablet, once-daily for 24 weeks
  Interventions: Drug: KRP-104
- Dose 4: KRP-104 20/120mg (Experimental): Tablet, once-daily for 24 weeks (dose switch from 20 to 120 mg at week 12)
  Interventions: Drug: KRP-104
- Placebo (Placebo Comparator): Tablet, once-daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KRP-104 — Tablet
  Arms: Dose 1: KRP-104 40 mg; Dose 2: KRP-104 80 mg; Dose 3: KRP-104 100 mg; Dose 4: KRP-104 20/120mg
Drug: Placebo — Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of KRP-104 on glycemic control in patients with type 2 diabetes inadequately controlled on metformin alone.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following criteria at the screening visit (Visit 1) will be eligible to participate in the trial:

1. Signed written informed consent;
2. Males and females 18 to 75 years of age, inclusive;
3. Females of childbearing potential must agree to use 2 adequate forms of barrier method contraception (eg, latex condom AND intrauterine device or a diaphragm) to avoid pregnancy while in the study;
4. On a stable dose (Greater than or equal to 10 weeks at the same dose) of metformin monotherapy (Less than or equal to 1500 mg/day or maximum tolerated dose), have an HbA1c greater than or equal to 7.0% and less than or equal to 10.5%; or

   * On metformin (less than or equal to 1500 mg/day) and 1 other antidiabetic agent (excluding TZD, insulin, or incretin therapies [DPP-4 inhibitors and GLP-1 analogues]) and have an HbA1c greater than or equal to 6.8% and less than or equal to 10.0%; or
   * Not on antidiabetic therapy (for at least 3 months prior to Visit 1) or have not been on a stable dose of metformin monotherapy for 10 weeks and have an HbA1c greater than or equal to 8.0% and less than or equal to 11.0%.

Exclusion Criteria:

1. History of type 1 diabetes mellitus or history of diabetic ketoacidosis or persistent hypoglycemia;
2. History or presence of alcoholism or drug abuse within the 2 years prior to dosing;
3. Typical consumption of greater than or equal to 10 drinks of alcohol weekly;
4. Presence of any of the following conditions:

   * Significant renal impairment (glomerular filtration rate less than 60 mL/min);
   * Diabetic gastroparesis;
   * Active liver disease (other than asymptomatic nonalcoholic fatty liver disease), cirrhosis, or symptomatic gallbladder disease;
5. Fasting plasma glucose/blood glucose greater than 240 mg/dL (13.3 mmol/L) at Visit 3 (Week -2) (1 laboratory retest permitted);
6. Body mass index less than or equal to 20 kg/m2 and greater than or equal to 48 kg/m2;
7. Systolic blood pressure <100 mmHg or >160 mmHg and diastolic blood pressure <50 mmHg or >100 mmHg at Visit 3 (Note: medication to control blood pressure is allowed and should be optimized and stabilized prior to Visit 3);
8. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 X the upper limit of normal (ULN) (1 laboratory retest permitted);
9. Creatine phosphokinase (CPK) greater than 2 X the ULN (if not explained by muscular trauma or exercise) (1 laboratory retest permitted);
10. Serum creatinine >1.5 mg/dL for males (132.6 μmol/L) and 1.4 mg/dL for females (123.8 μmol/L);
11. Fasting triglycerides (TG) >600 mg/dL (6.78 mmol/L) at Visit 3 (Week -2) (Note: diet/exercise and lipid-lowering medication to control elevated TG is allowed; medications should be optimized and stabilized prior to Visit 3);
12. Treatment with pioglitazone or rosiglitazone within the previous 10 weeks (Visit 1); treatment with incretin therapy (DPP-4 inhibitors or GLP-1 analogues) within the previous 4 weeks (Visit 1);
13. Treatment with any type of insulin (ie, injected or inhaled) within the previous 3 months;
14. Must meet other laboratory and Medical History clinical criteria. Please contact recruitment center for referrals

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2009-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diane J Plotkin, PhD, Study Director — ActivX Biosciences, Inc.
Locations (45):
- United States (17):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - Valley Village, California
  - Honolulu, Hawaii
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Delaware, Ohio
  - Marion, Ohio
  - Beaver, Pennsylvania
  - Jenkintown, Pennsylvania
  - Greer, South Carolina
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Sandy City, Utah
  - West Jordan, Utah
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Loma Hermos Buenos Aires
- Czechia (5):
  - Chrudim III
  - Holešov
  - Mělník
  - Ostrava
  - Prague
- Guatemala City, Guatemala
- Poland (6):
  - Bialystok
  - Gdansk
  - Krakow
  - Lodz
  - Warsaw
  - Wroclaw
- Russia (5):
  - Arkhangelsk
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Saint Petersburg
- South Africa (8):
  - Port Elizabeth, Eastern Cape
  - Bloemfontein, Free State
  - Johannesburg, Gauteng
  - Soweto, Gauteng
  - Durban, Kwazula-Natal
  - Cape Town, Western Cape
  - Paarl, Western Cape
  - Somerset West, Western Cape

REFERENCES:
- [Result] Plotkin DJ, Lewin A, Logan D, Kato T, Kozarich J, Wei X, Vest J, Orloff D. KRP-104, A Uniquely Prandial-Targeted DPP-4 Inhibitor. Abstract and Poster # 822, Presented at: European Association for the Study of Diabetes 38th Annual Meeting, Berlin Germany, October 1-5, 2012.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted in 55 medical clinics in 6 countries: US, Guatemala, South Africa, Russia, Czech Republic, Poland. First site opened 19 October 2009.
Pre-assignment Details: Variable screening duration to allow for wash-out of one oral therapy, optimization and stabilization of dose on metformin monotherapy (>= 10 weeks);followed by 2 week placebo run-in. Fasting CBG <240 mg/dL at start of run in and prior to randomization required.
Groups:
- Dose 1: KRP-104: 40 mg QD
- Dose 2: KRP-104: 80 mg QD
- Dose 3: KRP-104: 100 mg QD
- Dose 4: KRP-104: 20 mg /120 mg QD (dose switch at week12)
Period: Overall Study
Arm/Group | Placebo | Dose 1: KRP-104 | Dose 2: KRP-104 | Dose 3: KRP-104 | Dose 4: KRP-104
Started | 81 | 81 | 80 | 81 | 80
Completed | 70 | 74 | 73 | 76 | 75
Not Completed | 11 | 7 | 7 | 5 | 5
Not completed — Withdrawal by Subject | 4 | 2 | 1 | 3 | 1
Not completed — Adverse Event | 3 | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 2 | 2 | 2 | 1 | 0
Not completed — all other reasons combined | 2 | 2 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Dose 4: KRP-104: 20 mg QD (weeks 1-12)/120 mg QD (weeks 12-24)
- Total: Total of all reporting groups
Arm/Group | Placebo | Dose 1: KRP-104 | Dose 2: KRP-104 | Dose 3: KRP-104 | Dose 4: KRP-104 | Total
Number analyzed (Participants) | 81 | 81 | 80 | 81 | 80 | 403
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 69 | 66 | 64 | 73 | 332
  >=65 years | 21 | 12 | 14 | 17 | 7 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (9.43) | 54.2 (10.59) | 55.7 (9.10) | 56.3 (9.40) | 55.5 (8.27) | 55.8 (9.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 59 | 52 | 49 | 55 | 259
  Male | 37 | 22 | 28 | 32 | 25 | 144
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 21 | 21 | 20 | 103
  Czech Republic | 6 | 6 | 5 | 6 | 5 | 28
  Poland | 4 | 3 | 2 | 4 | 3 | 16
  Guatemala | 16 | 15 | 15 | 14 | 16 | 76
  South Africa | 21 | 23 | 23 | 22 | 22 | 111
  Russian Federation | 13 | 14 | 14 | 14 | 14 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline (Week 0) to Week 24
Description: Mean Change in HbA1c (%) from Baseline to Week 24 with LOCF, ITT population LS mean (SE)
Time Frame: Week 24
Population: Conducted analyses of ITT population of change in HbA1c from baseline (Week 0) to Week 24. If the Wk 24 measurement was missing, the last valid post-baseline observation (LOCF) algorithm was used to impute Week 24 value (1 on-treatment value required). Efficacy data collected after the initiation of rescue therapy was excluded from the analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: % HbA1c
Arm/Group | Placebo | Dose 1: KRP-104 | Dose 2: KRP-104 | Dose 3: KRP-104 | Dose 4: KRP-104
Number analyzed (Participants) | 78 | 79 | 79 | 80 | 79
% HbA1c | -0.09 (0.097) [-.28 to 0.10] | -0.41 (0) [-0.60 to -0.22] | -0.70 [-0.89 to -0.51] | -0.71 [-0.89 to -0.52] | -0.73 [-0.92 to -0.54]

2. Secondary Outcome: Change in Body Weight
Description: Mean Change in Body Weight (kg) from Baseline to Week 24 with LOCF- ITT
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: kg body weight on scale
Arm/Group | Placebo | Dose 1: KRP-104 | Dose 2: KRP-104 | Dose 3: KRP-104 | Dose 4: KRP-104
Number analyzed (Participants) | 78 | 79 | 79 | 80 | 79
kg body weight on scale | -0.73 (0.303) | -1.13 (0.303) | -1.31 (0.302) | -0.70 (0.300) | -0.18 (0.302)

3. Secondary Outcome: Percentage of Patients Achieving HbA1c Less Than 7%
Description: Subjects Achieving Target of Hemoglobin A1c <7.0% at Week 24 with LOCF - Intent-to-Treat Population
Time Frame: 24 weeks
Measure: Number; unit: % of subjects in group
Arm/Group | Placebo | Dose 1: KRP-104 | Dose 2: KRP-104 | Dose 3: KRP-104 | Dose 4: KRP-104
Number analyzed (Participants) | 78 | 79 | 79 | 80 | 79
% of subjects in group | 23.08 | 31.65 | 49.37 | 43.75 | 41.77

4. Secondary Outcome: Percentage of Patients Requiring Rescue Therapy for Elevated Glucose
Description: Percentage of Subjects Requiring Rescue Therapy - Intent-to-Treat Population
Time Frame: 24 weeks of treatment.
Measure: Number; unit: % of subjects in group
Arm/Group | Placebo | Dose 1: KRP-104 | Dose 2: KRP-104 | Dose 3: KRP-104 | Dose 4: KRP-104
Number analyzed (Participants) | 79 | 79 | 79 | 80 | 79
% of subjects in group | 6.33 | 10.1 | 5.06 | 3.75 | 3.8

ADVERSE EVENTS:
Time Frame: From first site open on 19 October 2009 through 30 days after last subject out on 20 January 2011, approximately 1 year 5 months.
Description: Only treatment related adverse events were reported in the clinical study report. There were no occurrences of serious adverse events that were considered related to drug, thus none met criterion of reportable event.
Arm/Group | Placebo | Dose 1: KRP-104 | Dose 2: KRP-104 | Dose 3: KRP-104 | Dose 4: KRP-104
Serious Adverse Events (participants affected / at risk) | 3/81 | 2/81 | 4/80 | 1/81 | 1/80
Other Adverse Events (participants affected / at risk) | 24/81 | 16/81 | 16/80 | 17/81 | 19/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Dose 1: KRP-104 (N=81) | Dose 2: KRP-104 (N=80) | Dose 3: KRP-104 (N=81) | Dose 4: KRP-104 (N=80)
Breast cancer (left breast) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — not related, start = study day 34
tuberculosis meningitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — not related, start date= study day 27 subject was subsequently also diagnosed with human immunodeficiency virus
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — study day 76, not related
Fracture Of The Left Anterior Lamina Papyracea (Ethmoid Bone) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — not related, start= day 35
Lyme Disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — not related, start= day 18
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — not related, start= day 86
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — not related, start = day 121
lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — not related, start= day 6
Cholecystolithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — not related, start=day 70
Intractable Low Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — not related, start= day 68
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — not related, start= day 119
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Dose 1: KRP-104 (N=81) | Dose 2: KRP-104 (N=80) | Dose 3: KRP-104 (N=81) | Dose 4: KRP-104 (N=80)
Urinary tract infection (Infections and infestations) | 5 | 6 | 9 | 5 | 6
Influenza (Infections and infestations) | 5 | 4 | 2 | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 1 | 2 | 4
Diarrhea (Gastrointestinal disorders) | 4 | 1 | 2 | 5 | 2
Hypertension (Vascular disorders) | 6 | 2 | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No explicit limitations on discussion by PI. PI may not publish results before a coordinated multicenter publication has been submitted for publication, marketing approval obtained, or until 7 years after the study has ended, whichever occurs first. Thereafter, the study site will have the opportunity to publish the results of the study, provided that the Sponsor has had the opportunity to review and comment on the study site's proposed publication prior to it being submitted for publication.